CLINICAL TRIAL: NCT03078478
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec and Insulin Glargine 300 Units/mL in Subjects With Type 2 Diabetes Mellitus Inadequately Treated With Basal Insulin With or Without Oral Antidiabetic Drugs
Acronym: CONCLUDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-4252; U1111-1184-8175 (Other: WHO); 2016-002801-20 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-03-13 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDeg 200 U/mL (Experimental)
  Interventions: Drug: Insulin degludec
- IGlar 300 U/mL (Active Comparator)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin degludec — For subcutaneous (s.c., under the skin) injection once daily
  Arms: IDeg 200 U/mL
Drug: Insulin glargine — For subcutaneous (s.c., under the skin) injection once daily
  Arms: IGlar 300 U/mL

SUMMARY:
This trial is conducted in Europe and North America. The aim of the trial is to compare the efficacy and safety of insulin degludec and insulin glargine 300 units/mL in subjects with type 2 diabetes mellitus inadequately treated with basal insulin with or without oral antidiabetic drugs. Due to change in glycaemic data collection process, this trial is amended to allow for a full 36 weeks (maintenance 2 period) of the use of the new process.

ELIGIBILITY:
Inclusion criteria: - Male or female, age above or equal to 18 years at the time of signing informed consent. - Subjects fulfilling at least one of the below criteria (For this inclusion criterion the aim is to include minimum 80% of individuals with a previous episode of hypoglycaemia (criterion e). The remaining subjects will have to fulfil at least one of criteria a-d.): - a) Experienced at least one severe hypoglycaemic episode within the last year (according to the ADA definition, April 2013 (An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.). - b) Moderate chronic renal failure, defined as glomerular filtration rate 30 - 59 mL/min/1.73 m^2 per CKD-EPI by central laboratory analysis. - c) Hypoglycaemic symptom unawareness (History of impaired autonomic responses (tremulousness, sweating, palpitations, and hunger) during hypoglycaemia). - d) Treated with insulin for more than 5 years. - e) Episode of hypoglycaemia (defined by symptoms of hypoglycaemia and/or episode with low glucose measurement (equal to or below 70 mg/dL [equal to or below 3.9 mmol/L])) within the last 12 weeks prior to Visit 1 (screening). - Subjects diagnosed (clinically) with type 2 diabetes mellitus. - Treated with basal only insulin (once daily or twice-daily insulin (insulin detemir; insulin glargine 100 U/mL, biosimilar of insulin glargine 100 U/mL or insulin Neutral Protamine Hagedorn)) equal to or above 90 days prior to the day of screening with or without any of the following anti-diabetic drugs with stable doses for equal to or above 90 days prior to screening: - a) Metformin - b) Dipeptidyl peptidase -4 inhibitor - c) Sodium-glucose co-transporter 2 inhibitor - d) Alpha-glucosidase-inhibitors (acarbose) - e) Thiazolidinediones - f) Marketed oral combination products only including the products listed in criteria 5a-5e - HbA1c equal to or below 9.5% (80 mmol/mol) at screening by central laboratory analysis. - BMI equal to or below 45 kg/m^2. Exclusion Criteria: - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (195):
- United States (138):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Fountain Hills, Arizona
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Downey, California
  - Novo Nordisk Investigational Site, Duarte, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Moreno Valley, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Pomona, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Stanford, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, West Hills, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Englewood, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Brandon, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Springs, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Ormond Beach, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Wauconda, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Mishawaka, Indiana
  - Novo Nordisk Investigational Site, Valparaiso, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Bloomfield Hills, Michigan
  - Novo Nordisk Investigational Site, Richfield, Minnesota
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Kalispell, Montana
  - Novo Nordisk Investigational Site, Elkhorn, Nebraska
  - Novo Nordisk Investigational Site, Fremont, Nebraska
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, East Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, West Columbia, South Carolina
  - Novo Nordisk Investigational Site, Dakota Dunes, South Dakota
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Kerrville, Texas
  - Novo Nordisk Investigational Site, New Braunfels, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Bennington, Vermont
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
  - Novo Nordisk Investigational Site, West Allis, Wisconsin
- Canada (9):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Markham, Ontario
  - Novo Nordisk Investigational Site, Oakville, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
- Denmark (6):
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Estonia (3):
  - Novo Nordisk Investigational Site, Pärnu
  - Novo Nordisk Investigational Site, Tallinn
  - Novo Nordisk Investigational Site, Viljandi
- Germany (10):
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Lingen
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- Greece (4):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Nikaia
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Szombathely
- Norway (5):
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Hoenefoss
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Skedsmokorset
  - Novo Nordisk Investigational Site, Trondheim
- Poland (7):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Manatí
  - Novo Nordisk Investigational Site, Ponce
- Romania (4):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Buzău
  - Novo Nordisk Investigational Site, Galati
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Background] Philis-Tsimikas A, Stratton I, Norgard Troelsen L, Anker Bak B, Leiter LA. Efficacy and Safety of Degludec Compared to Glargine 300 Units/mL in Insulin-Experienced Patients With Type 2 Diabetes: Trial Protocol Amendment (NCT03078478). J Diabetes Sci Technol. 2019 May;13(3):498-506. doi: 10.1177/1932296819841585. Epub 2019 Apr 11. PMID 30974986
- [Result] Philis-Tsimikas A, Klonoff DC, Khunti K, Bajaj HS, Leiter LA, Hansen MV, Troelsen LN, Ladelund S, Heller S, Pieber TR; CONCLUDE Study Group. Risk of hypoglycaemia with insulin degludec versus insulin glargine U300 in insulin-treated patients with type 2 diabetes: the randomised, head-to-head CONCLUDE trial. Diabetologia. 2020 Apr;63(4):698-710. doi: 10.1007/s00125-019-05080-9. Epub 2020 Jan 27. PMID 31984443
- [Derived] Evans M, Moes RGJ, Pedersen KS, Gundgaard J, Pieber TR. Cost-Effectiveness of Insulin Degludec Versus Insulin Glargine U300 in the Netherlands: Evidence From a Randomised Controlled Trial. Adv Ther. 2020 May;37(5):2413-2426. doi: 10.1007/s12325-020-01332-y. Epub 2020 Apr 18. PMID 32306247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 230 sites in 11 countries as follows. Number of sites that screened and randomised participants to treatment are given in parenthesis. Canada:(9/9), Denmark: (6/6), Estonia: (5/5), Germany: (11 /11), Greece: (7/7), Hungary: (9/9), Norway: (4/4), Poland: (9/9), Romania: (5/4), Serbia: (8/8), United States: (157/153).
Pre-assignment Details: The participants were previously treated with basal insulin once daily or twice daily ± oral anti-diabetic drugs excluding sulfonylureas/glinides. Pre-trial insulin was discontinued and the subjects continued their pre-trial oral anti-diabetic drugs (OADs).
Groups:
- Insulin Degludec U200: Participants received insulin degludec 200 units/mL once daily as subcutaneous injections (in the thigh, upper arm or abdomen) ± oral anti-diabetic drugs. The daily basal insulin dose was reduced by 20% from their pre-trial dose. Insulin dose was adjusted once weekly by the investigator, based on the mean of three fasting self measured plasma glucose (SMPG) values, to reach a SMPG of 4.0-5.0 mmol/L (71-90 mg/dL). The treatment duration was up to 88 weeks divided into; a 16-week titration period, an up to 36-week maintenance period 1 (variable length) and a 36-week maintenance period 2.
- Insulin Glargine U300: Participants received insulin glargine 300 units/mL once daily as subcutaneous injections (in the thigh, upper arm or abdomen) ± pre-trial oral anti-diabetic drugs. The dose of IGlar U300 corresponded to the pre-trial daily basal insulin dose. Insulin dose was adjusted once weekly by the investigator, based on the mean of three fasting SMPG values, to reach a SMPG of 4.0-5.0 mmol/L (71-90 mg/dL). The treatment duration was up to 88 weeks divided into; a 16-week titration period, an up to 36-week maintenance period 1 (variable length) and a 36-week maintenance period 2.
Period: Titration Period (16 Weeks)
Arm/Group | Insulin Degludec U200 | Insulin Glargine U300
Started | 805 | 804
Full Analysis Set | 805 | 804
Safety Analysis Set | 802 | 798
Completed | 805 | 804
Not Completed | 0 | 0
Period: Maintenance Period 1 (36 Weeks)
Arm/Group | Insulin Degludec U200 | Insulin Glargine U300
Started | 805 | 804
Completed | 758 | 761
Not Completed | 47 | 43
Not completed — Withdrawal by Subject | 36 | 36
Not completed — Lost to Follow-up | 7 | 4
Not completed — Death | 3 | 3
Not completed — Subject withdrawal reason not collected | 1 | 0
Period: Maintencance Period 2 (36 Weeks)
Arm/Group | Insulin Degludec U200 | Insulin Glargine U300
Started | 758 | 761
Completed | 733 | 734
Not Completed | 25 | 27
Not completed — Withdrawal by Subject | 18 | 13
Not completed — Lost to Follow-up | 3 | 6
Not completed — Death | 4 | 6
Not completed — Not reconsenting | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec U200 | Insulin Glargine U300 | Total
Number analyzed (Participants) | 805 | 804 | 1609
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (10) | 62.8 (10) | 62.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333 | 368 | 701
  Male | 472 | 436 | 908
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 100 | 184
  Not Hispanic or Latino | 721 | 704 | 1425
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 25 | 29 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 78 | 65 | 143
  White | 693 | 699 | 1392
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes During Maintenance 2 (36 Weeks)
Description: Severe or BG confirmed symptomatic hypoglycaemia was evaluated during maintenance 2 (36 weeks) period. Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA 2013 classification or blood glucose (BG) confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe or BG-confirmed symptomatic hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 36 Weeks
Population: The safety analysis set (SAS) comprised all subjects who received at least one dose of the investigational product or comparator.
Measure: Number; unit: Episodes/(PYE*100)
Groups:
- Insulin Degludec 200: Participants received insulin degludec 200 units/mL once daily as subcutaneous injections (in the thigh, upper arm or abdomen) ± oral anti-diabetic drugs. The daily basal insulin dose was reduced by 20% from their pre-trial dose. Insulin dose was adjusted once weekly by the investigator, based on the mean of three fasting self measured plasma glucose (SMPG) values, to reach a SMPG of 4.0-5.0 mmol/L (71-90 mg/dL). The treatment duration was up to 88 weeks divided into; a 16-week titration period, an up to 36-week maintenance period 1 (variable length) and a 36-week maintenance period 2.
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 742 | 741
Episodes/(PYE*100) | 216.8 | 243.9
Statistical Analysis 1: Comparison: Insulin Degludec 200 vs Insulin Glargine U300; The number of episodes is analysed using a negative binomial regression model (log link) with the logarithm of the time period in which a hypoglycaemic episode was considered treatment emergent as offset. The model includes treatment, number of OADs, region, sex and dosing time as fixed factors, and age as a covariate. Missing values are imputed through multiple imputation by treatment arm, based on a Poisson model; Test type: Superiority; p = 0.1715, Regression, Cox; Treatment rate ratio = 0.88, 95% CI 2-sided [0.73 to 1.06]

2. Secondary Outcome: Basal Insulin Dose (U) at End of Treatment (up to 88 Weeks)
Description: The observed mean daily basal insulin doses was evaluated at the end of trial (88 weeks).
Time Frame: 88 weeks
Population: The safety analysis set (SAS) comprised all subjects who received at least one dose of the investigational product or comparator. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 703 | 704
Units | 66.6 (48.54) | 73.0 (48.48)

3. Secondary Outcome: Number of Nocturnal, Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes During Maintenance 2 (36 Weeks)
Description: Nocturnal severe or BG confirmed symptomatic hypoglycaemia was evaluated during maintenance 2 (36 weeks). The nocturnal period defined as the period between 00:01 and 05:59 a.m. (both inclusive). Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA 2013 classification or blood glucose (BG) confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe or BG-confirmed symptomatic hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 36 weeks
Population: as for outcome 2
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 742 | 741
Episodes/(PYE*100) | 62.30 | 93.75

4. Secondary Outcome: Number of Severe Hypoglycaemic Episodes During Maintenance 2 (36 Weeks)
Description: Severe hypoglycaemia are those episodes positively adjudicated by the event adjudication committee according to the ADA definition of a severe hypoglycaemic episode. This was evaluated for maintenance 2 period. The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 36 weeks (maintenance 2)
Population: as for outcome 2
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 742 | 741
Episodes/(PYE*100) | 0.98 | 4.88

5. Secondary Outcome: Change in HbA1c From Baseline to End of Treatment (up to 88 Weeks)
Description: Change in glycosylated haemoglobin (HbA1c) was evaluated from baseline to end of treatment period (week 88).
Time Frame: Week 0, week 88
Population: The full analysis set (FAS) comprised all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 694 | 700
Percentage of HbA1c | -0.54 (0.91) | -0.46 (0.90)

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to End of Treatment (up to 88 Weeks)
Description: Change in fasting plasma glucose (FPG) was evaluated from baseline to end of treatment period (week 88).
Time Frame: Week 0, week 88
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 685 | 689
mg/dL | -35.50 (49.34) | -25.68 (56.69)

7. Secondary Outcome: Percentage of Participants With FPG ≤ 7.2 mmol/L (130 mg/dL) at End of Treatment (up to 88 Weeks) (Yes/no)
Description: Participants achieving a fasting plasma glucose value of less than or equal to 7.2 mmol/L (130 mg/dL) at end of treatment (up to 88 weeks).
Time Frame: At 88 weeks
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 701 | 700
Percentage of participants
  Yes | 84.0 | 72.0
  No | 16.0 | 28.0

8. Secondary Outcome: Percentage of Participants With FPG ≤ 5.0 mmol/L (90 mg/dL) at End of Treatment (up to 88 Weeks) (Yes/no)
Description: Participants achieving a fasting plasma glucose value of less than or equal to 5.0 mmol/L (90 mg/dL) at end of treatment (up to 88 weeks).
Time Frame: At 88 weeks
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 701 | 700
Percentage of participants
  Yes | 31.5 | 21.7
  No | 68.5 | 78.3

9. Secondary Outcome: Percentage of Participants With HbA1c < 7.0% (53 mmol/Mol) at End of Treatment (up to 88 Weeks) and no Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During Maintenance 2 (36 Weeks) (Yes/no)
Description: Participants achieving target HbA1c of less than 7.0% at the end of treatment (88 weeks) without severe or BG-confirmed hypoglycaemia during maintenance 2 (36 weeks).
Time Frame: End of Treatment (up to 88 Weeks)
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 694 | 700
Percentage of participants
  Yes | 35.3 | 30.0
  No | 64.7 | 70.0

10. Secondary Outcome: Percentage of Participants With HbA1c < 7.0% (53 mmol/Mol) at End of Treatment (up to 88 Weeks) and no Nocturnal, Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes During Maintenance 2 (36 Weeks) (Yes/no)
Description: Participants achieving target HbA1c of less than 7.0% at the end of treatment (88 weeks) without nocturnal severe or BG-confirmed hypoglycaemia during maintenance 2 (36 weeks).
Time Frame: At 88 weeks
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 694 | 700
Percentage of participants
  Yes | 47.4 | 39.3
  No | 52.6 | 60.7

11. Secondary Outcome: Change in Mean Pre-breakfast Self-measured Plasma Glucose Used for Titration From Baseline to End of Treatment (up to 88 Weeks)
Description: Participants measured their pre-breakfast self-measured plasma glucose (SMPG) value until end of treatment (week 88). Mean pre-breakfast self-measured plasma glucose used for titration at baseline and end of treatment (up to 88 weeks) are presented.
Time Frame: Week 0, week 88
Population: Full analysis set (FAS) included all randomised subjects. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 805 | 804
mmol/L
  Baseline (week 0): number analyzed (Participants) | 329 | 349
  Baseline (week 0) | 8.39 (2.73) | 8.41 (2.75)
  End of treatment (week 88): number analyzed (Participants) | 690 | 694
  End of treatment (week 88) | 5.46 (1.08) | 5.56 (1.23)

12. Secondary Outcome: Number of Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes During Treatment (up to 88 Weeks)
Description: Severe or BG confirmed symptomatic hypoglycaemia was evaluated during treatment (up to 88 weeks). Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA 2013 classification or blood glucose (BG) confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe or BG-confirmed symptomatic hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 88 weeks
Population: as for outcome 1
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 802 | 798
Episodes/(PYE*100) | 137.8 | 163.7

13. Secondary Outcome: Number of Nocturnal, Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes During Treatment (up to 88 Weeks)
Description: Nocturnal severe or BG confirmed symptomatic hypoglycaemia was evaluated at the end of trial (88 weeks). The nocturnal period defined as the period between 00:01 and 05:59 a.m. (both inclusive). Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA 2013 classification or blood glucose (BG) confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe or BG-confirmed symptomatic hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 88 weeks
Population: as for outcome 1
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 802 | 798
Episodes/(PYE*100) | 36.93 | 60.03

14. Secondary Outcome: Number of Severe Hypoglycaemic Episodes During Treatment (up to 88 Weeks)
Description: Severe hypoglycaemia are those episodes positively adjudicated by the event adjudication committee according to the ADA definition of a severe hypoglycaemic episode. This was evaluated for the total trial period (88 weeks). The observed rates (number of episodes divided by patient years of exposure multiplied by 100) of severe hypoglycaemic episodes per patient years of exposure (PYE) is presented in this endpoint results.
Time Frame: 88 weeks
Population: as for outcome 1
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 802 | 798
Episodes/(PYE*100) | 2.06 | 5.21

15. Secondary Outcome: Number of Adverse Events From Randomisation to End of Maintenance Period 2 (up to 88 Weeks)
Description: The adverse events presented are treatment emergent. A treatment-emergent AE (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last days of randomised treatment or had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last date of randomised treatment. Number of adverse events expressed in rates, from randomisation to end of maintenance period 2 (up to 88 weeks) is presented. Rate = number of events divided by patient years of exposure multiplied by 100.
Time Frame: 88 weeks
Population: as for outcome 1
Measure: Number; unit: Episodes/(PYE*100)
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 802 | 798
Episodes/(PYE*100) | 367.32 | 365.42

16. Secondary Outcome: Change in Body Weight From Baseline to End of Treatment (up to 88 Weeks)
Description: Change in body weight, measured in kilograms, from baseline (week 0) to end of treatment (week 88).
Time Frame: Week 0, week 88
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Degludec 200 | Insulin Glargine U300
Number analyzed (Participants) | 701 | 703
kg | 2.9 (5.17) | 1.7 (5.84)

ADVERSE EVENTS:
Time Frame: From the first trial-related activity after the subject had signed the informed consent until the End of Trial (week 88) + 7 days follow-up period. Results are based on the safety analysis set (SAS), which comprised all participants who received at least one dose of trial product.
Description: A treatment-emergent AE (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last days of randomised treatment or had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last date of randomised treatment.
Groups:
- IDeg U200: Participants received insulin degludec 200 units/mL once daily as subcutaneous injections (in the thigh, upper arm or abdomen) ± oral anti-diabetic drugs. The daily basal insulin dose was reduced by 20% from their pre-trial dose. Insulin dose was adjusted once weekly by the investigator, based on the mean of three fasting SMPG values, to reach a SMPG of 4.0-5.0 mmol/L (71-90 mg/dL). The treatment duration was up to 88 weeks divided into; a 16-week titration period, an up to 36-week maintenance period 1 (variable length) and a 36-week maintenance period 2.
- IGlar U300: Participants received insulin glargine 300 units/mL once daily as subcutaneous injections (in the thigh, upper arm or abdomen) ± pre-trial oral anti-diabetic drugs. The dose of IGlar U300 corresponded to the pre-trial daily basal insulin dose. Insulin dose was adjusted once weekly by the investigator, based on the mean of three fasting SMPG values, to reach a SMPG of 4.0-5.0 mmol/L (71-90 mg/dL). The treatment duration was up to 88 weeks divided into; a 16-week titration period, an up to 36-week maintenance period 1 (variable length) and a 36-week maintenance period 2.
Arm/Group | IDeg U200 | IGlar U300
All-Cause Mortality (participants affected / at risk) | 7/802 | 9/798
Serious Adverse Events (participants affected / at risk) | 167/802 | 141/798
Other Adverse Events (participants affected / at risk) | 496/802 | 476/798
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg U200 (N=802) | IGlar U300 (N=798)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 8 (9)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 2 (2)
Angina unstable (Cardiac disorders) | 6 (7) | 4 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 5 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Capsular contracture associated with breast implant (General disorders) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (3) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 10 (10) | 5 (5)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 3 (3) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (4)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drug administered in wrong device (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Eye haematoma (Eye disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenterostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (8) | 19 (21)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 3 (4) | 9 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Intentional product misuse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 4 (4)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Multiple drug therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 2 (2)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (3) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parametritis (Infections and infestations) | 0 (0) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 6 (8) | 9 (9)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 2 (2)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 5 (5)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vitreous adhesions (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg U200 (N=802) | IGlar U300 (N=798)
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 (59) | 65 (84)
Back pain (Musculoskeletal and connective tissue disorders) | 59 (73) | 62 (70)
Bronchitis (Infections and infestations) | 48 (54) | 46 (46)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (60) | 46 (53)
Diarrhoea (Gastrointestinal disorders) | 72 (90) | 79 (97)
Headache (Nervous system disorders) | 51 (61) | 62 (70)
Influenza (Infections and infestations) | 59 (64) | 41 (44)
Nasopharyngitis (Infections and infestations) | 152 (253) | 161 (265)
Nausea (Gastrointestinal disorders) | 43 (53) | 50 (56)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 (49) | 43 (49)
Sinusitis (Infections and infestations) | 45 (58) | 40 (53)
Upper respiratory tract infection (Infections and infestations) | 145 (199) | 122 (177)
Urinary tract infection (Infections and infestations) | 49 (58) | 47 (65)
Vomiting (Gastrointestinal disorders) | 26 (30) | 40 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT03078478/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03078478/SAP_001.pdf